CLINICAL TRIAL: NCT06335394
Title: A Prospective Multicentre Single-arm Study in Adults to Evaluate the Safety and Preliminary Efficacy of the Autologous 3D Osteogenic Implant NVD-003 for Bone Reconstruction for the Treatment of Recalcitrant Lower Limb Nonunion
Brief Title: Prospective Study in Adults Evaluating Safety & Efficacy of NVD003 for Bone Reconstruction to Treat Lower Limb Nonunion
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novadip Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NVD003-CLN01
Record Dates: First submitted 2023-11-21; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Recalcitrant Lower Limb Nonunion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-arm study (Experimental): NVD003
  Interventions: Other: NVD003

INTERVENTIONS:
Other: NVD003 — Autologous osteogenic implant NVD-003 for bone reconstruction

SUMMARY:
The goal of this clinical trial is to evaluate the safety and preliminary efficacy of the autologous 3D osteogenic implant NVD-003 for bone reconstruction for the treatment of recalcitrant lower limb nonunion.

DETAILED DESCRIPTION:
This is a first in man study conducted as a prospective, single-arm, non-randomized clinical study. A sample of 5 to 10 patients will be enrolled in the study in order to assess the safety of the use of NVD-003 bone graft implantation in patients with recalcitrant lower limb nonunion.

The sample size of 5 to 10 patients was considered sufficient to give a preliminary indication on the safety of the ATMP.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adult subject (≥18 years).
2. Radiographic images not older than 3 months, confirming lower limb nonunion, defined as the absence of clinical and radiographic progression towards healing over 3 consecutive months on serial radiographs and minimum 9 months after the first attempt of surgical bone repair, or minimum 6 months after the second (or any subsequent) attempt of surgical bone repair.
3. Radiologic single, meta- and/or diaphyseal bone defect with a maximum size of 4 cm (in case of a void that does not transverse the whole width of the bone, the total volume cannot exceed the volume corresponding to the 4 cm gap).
4. The impaired limb is salvageable, and the patient is eligible for the intended surgical procedure according to the standard hospital practice.
5. Documented normal or low bone density: Bone density scan determined by Dual Energy X-Ray Absorptiometry DEXA scan on lumbar spine and hip (bone mineral density T-scores above -2.5). An examination ≤ 1-year-old before screening is acceptable.
6. The subject is, in the Investigator's opinion, psychosocially, mentally, and physically able to fully comply with this protocol, including the postoperative regimen and follow-up visits.
7. Use of an effective birth control method for 2 months prior to the date of the intended surgical intervention up to Visit V7 for women of childbearing potential.
8. Negative urinary pregnancy test for women of childbearing potential.
9. At screening, safety local laboratory test results are medically acceptable to undergo surgery (see Section 7.3.2) and serology results are in accordance with country specific requirements for donation of Human Body Material.
10. At time of adipose tissue collection, central laboratory serology and molecular tests panel for Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), and syphilis are in accordance with Belgian specific requirements for release of Human Body Material.
11. The subject has understood the nature of the study, agrees to its provisions, and has accepted to participate in the study and to follow all study procedures. This is acknowledged by signing the informed consent as approved by the required Institutional Review Board/Ethics Committee and the national competent authorities.
12. Patient fulfils the criteria to donate his human body material (adipose tissue) and is suitable to undergo a liposuction.

Exclusion Criteria:

1. The subject has a Body Mass Index (BMI) ≤ 20 kg/m² or ≥ 40 kg/m², or of ≥35 kg/m² with obesity-related health conditions, such as high blood pressure or diabetes.
2. Multifocal or comminuted fractures.
3. A planned use of an external fixator is not allowed as of the grafting surgery (V1) until V7.
4. Documented osteoporosis: bone density determined using DEXA scan on lumbar spine and hip: bone mineral density T-scores of -2.5 and below. An examination ≤ 1-year-old before screening is acceptable.
5. Pregnant or breast-feeding woman.
6. The subject shows signs of an active drug or alcohol dependence, serious current illness, mental illness or any other factors which, in the opinion of the investigator, will interfere with study conduct or the interpretation of the results.
7. The patient has a history of solid organ transplant at any point in the past or is on the waiting list for future organ transplantation.
8. The subject previously received a cellular therapy treatment at any point in time (as per protocol description).
9. Previous exposure to any experimental therapy with another investigational drug within 60 days prior to screening or enrolment in any concurrent study that may confound the results of this study.
10. Any signs or suspicion of an active local (area of the future surgical site), or systemic infection before the induced membrane surgery or the grafting surgery.
11. Known allergy to any antibiotics commonly used to treat Staphylococcus aureus (including methicillin-resistant Staphylococcus aureus) or coagulase-negative staphylococci.
12. Diagnosis of HIV, HBV (HBsAg or PCR positive), HCV, Human T-cell Lymphotropic Virus (HTLV) 1 or 2, or syphilis infection (as confirmed by serology and nucleic acid test (NAT) by Tissue Establishment).
13. Chronic use of immunosuppressive therapy (immunosuppressant/ immunotherapy) due to inflammatory or systemic disease.
14. Any clinically relevant chronic disease associated with renal or hepatic insufficiency or any chronic disease of such severity that surgery could be detrimental to the survival of the patient.
15. Subjects with poorly controlled diabetes mellitus type 2 as assessed by glycated haemoglobin (HbA1C) ≥ 10%.
16. Subjects with poorly controlled thyroid diseases (unstable despite proper medication).
17. Subjects with documented metabolic bone disease (based on the investigator judgment) such as, but not limited to, osteogenesis imperfecta or osteomalacia.
18. Chronic, current or planned during study use of any medications that might affect bone metabolism or the quality of bone formation such as, but not limited to, bisphosphonates, steroids, methotrexate, anticoagulant therapies, immunosuppressant therapy or immunotherapy. However, short lasting surgery-related prophylactic treatments such as antibiotics, analgesics and low molecular heparin drugs may be administered according to hospital recommendations.
19. Existing malignant tumour in the vicinity of the graft or a resected one not cured for more than 5 years.
20. Any other illness which might reduce life expectancy to less than 2 years from screening.
21. The subject is a prisoner.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-08-02 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2028-05-15 (Estimated)

PRIMARY OUTCOMES:
Safety - Adverse Events | From graft implantation until completion of visit 24 months
  All Adverse Events (AEs) including Serious Adverse Events (SAEs), Adverse Events of Special Interest (AESI) and Procedure Related AE's (PRAE).
Safety - Abnormalities of vital signs | At hospital discharge (1-2 weeks after grafting surgery), at visit 1,5 months, at visit 3 months, at visit 6 months, at visit 12 months and visit 24 months
  Vital signs abnormalities: blood pressure
Safety - Abnormalities of vital signs | At hospital discharge (1-2 weeks after grafting surgery), at visit 1,5 months, at visit 3 months, at visit 6 months, at visit 12 months and visit 24 months
  Vital signs abnormalities: heart rate
Safety - Abnormalities of physical examination | At hospital discharge (1-2 weeks after grafting surgery), at visit 1,5 months, at visit 3 months, at visit 6 months, at visit 12 months and visit 24 months
  Physical examinations abnormalities: cardiovascular system
Safety - Abnormalities of physical examination | At hospital discharge (1-2 weeks after grafting surgery), at visit 1,5 months, at visit 3 months, at visit 6 months, at visit 12 months and visit 24 months
  Physical examinations abnormalities: respiratory system
Safety - Abnormalities of physical examination | At hospital discharge (1-2 weeks after grafting surgery), at visit 1,5 months, at visit 3 months, at visit 6 months, at visit 12 months and visit 24 months
  Physical examinations abnormalities: legs examination (inspection of both legs and extensive examination of the affected leg)
Safety - Abnormalities of laboratories | At hospital discharge (1-2 weeks after grafting surgery), at visit 1,5 months, at visit 3 months, at visit 6 months, at visit 12 months and visit 24 months
  Safety laboratories abnormalities: blood sampling: haematology (tests that yield information on the qualitative and quantitative composition of the cellular components of the blood)
Safety - Abnormalities of laboratories | At hospital discharge (1-2 weeks after grafting surgery), at visit 1,5 months, at visit 3 months, at visit 6 months, at visit 12 months and visit 24 months
  Safety laboratories abnormalities: blood sampling: coagulation (measure your blood's ability to clot, and how long it takes to clot)
Safety - Abnormalities of laboratories | At hospital discharge (1-2 weeks after grafting surgery), at visit 1,5 months, at visit 3 months, at visit 6 months, at visit 12 months and visit 24 months
  Safety laboratories abnormalities: blood sampling: biochemistry (tests to evaluate organ function, electrolyte status, hormone levels and more (calcium, vitamin D))

SECONDARY OUTCOMES:
Healing efficacy: plain X-ray | At 6 weeks, 3 months, 6 months, 12 months, at additional visits (if no healing at 12 months after graft implant surgery) up to 24 months.
  Plain X-ray healing defined as 3 united cortices (the strong type of bone on the outer layer) out of 4, on antero-posterior and lateral X-ray views
Healing efficacy: CT-scan | At 6, 12 and 24 months
  Computerized Tomography (CT)-scan healing defined as 3 united cortices out of 4
Healing efficacy: average time from Investigational Medicinal Product grafting surgery till first observation of plain X-ray and CT-scan confirmed fracture healing | Average time from IMP grafting surgery till first observation of plain X-ray and CT-scan up to 24 months
  The average time from IMP grafting surgery till first observation of plain X-ray and CT-scan confirmed fracture healing
Healing efficacy: investigator assessed clinical healing | From 6 weeks post-grafting onwards up to 24 months
  Investigator assessed clinical healing based on the overall clinical evaluation of the patient: ability to bear weight (non-weight bearing, toe-touch weight bearing, partial weight bearing, full weight bearing and full weight bearing with walking), the pain score at palpation at the fracture site (patient to rate the pain from 0 to 10 with the understanding that 0 is equal to no pain and 10 is equal to worst possible pain) and the pain medication intake by the patient.
Healing efficacy: average time from IMP grafting surgery to Investigator assessed clinical healing | Time from grafting surgery till first observation of investigator assessed clinical healing up to 24 months
  The average time from IMP grafting surgery to Investigator assessed clinical healing
Grafting Surgery parameters | Duration of grafting surgery (visit 1) and duration of hospitalization after grafting surgery (visit 2)
  Parameter 1: duration of grafting surgery
Grafting Surgery parameters | Duration of grafting surgery (visit 1) and duration of hospitalization after grafting surgery (visit 2)
  Parameter 2: duration of hospitalization
Complications: rate of subsequent surgical interventions | At 12 and 24 months post-implant surgery
  Rate of subsequent surgical interventions (e.g. revision, removal, reoperation and/or supplemental fixation)
Quality of Life: pain evaluation | At screening and at 6 weeks, 3, 6, 12 and 24 months post-graft
  Pain evaluation with the Brief Pain Inventory (Short Form) (BPI-SF) (pain severity and pain interference with function)
Quality of Life: questionnaire EuroQol-5 Dimensions | At screening and at 6 weeks, 3, 6, 12 and 24 months post-graft
  QoL questionnaire EuroQol-5 Dimensions (EQ-5D-5L)
Quality of Life: overall treatment effect | At 3, 6, 12 and 24 months post-graft
  Overall Treatment Effect rating scale
General Pre-graft implantation safety: all SAEs, AESI and PRAE | Pre-graft implantation
  All AEs including Serious Adverse Events (SAEs), Adverse Events of Special Interest (AESI) and Procedure Related AE's (PRAE).
All SAEs during the extended safety follow-up period | During the extended safety follow-up period (between 24 months FU visit and 5 years post-grafting surgery)
  All Serious Adverse Events (SAEs).

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Marchal, MD, Principal Investigator — CHU Ambroise Paré
Locations (10):
- Belgium (8):
  - Centre Hospitalier Interregional Edith Cavel (CHIREC) - Clinique Ste Anne-St Remi, Anderlecht
  - Algemeen Ziekenhuis (AZ) Sint-Jan Brugge - Oostende AV - Campus Sint-Jan, Bruges
  - Centre Hospitalier Universitaire CHU/UVC Brugmann (Site Horta), Brussels
  - Grand Hôpital De Charleroi, Charleroi
  - Ziekenhuis Oost-Limburg (ZOL), Genk
  - Universitair Ziekenhuis Leuven, Campus Gasthuisberg, Leuven
  - CHU Ambroise Paré, Mons
  - Centre Hospitalier Regional De Namur, Namur
- Centre Hospitalier de Luxembourg, Luxembourg, Luxembourg
- University Hospital Basel, Basel, Switzerland